CLINICAL TRIAL: NCT00776100
Title: A Randomized Phase II Study of Oligometastatic Stage IV Non-Small Cell Lung Cancer (NSCLC) Treated With Systemic Therapy Plus Either Radiotherapy to All Sites of Gross Residual Disease or No Radiotherapy
Brief Title: Radiation Therapy or Observation After Chemotherapy in Treating Patients With Stage IV Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated prematurely due to slow accrual.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0724; NCI-2009-00664 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000616868 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer; adenosquamous cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Watchful Waiting; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Other): Patients undergo observation for 6 weeks.
  Interventions: Other: clinical observation
- Arm II (Experimental): Patients undergo radiotherapy 5 days a week for 6 weeks to all sites of gross disease.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Other: clinical observation — Patients undergo observation for 6 weeks.
  Arms: Arm I
Radiation: radiation therapy — Patients undergo radiotherapy 5 days a week for 6 weeks.
  Arms: Arm II

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Sometimes, after chemotherapy, the tumor may not need more treatment until it progresses. In this case, observation may be sufficient. It is not yet known whether radiation therapy is more effective than observation after chemotherapy in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying how well radiation therapy works compared with observation after chemotherapy in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether the addition of radiotherapy to radiographically apparent residual disease after an initial course of standard chemotherapy results in an improvement in overall survival of patients with oligometastatic stage IV non-small cell lung cancer.

Secondary

* To compare the progression-free survival of patients treated with radiotherapy vs observation after standard chemotherapy.
* To compare the time to disease progression and time to treatment failure in these patients.
* To compare the confirmed response rate in these patients.
* To compare the duration of response in these patients.
* To compare the adverse events in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior treatment with bevacizumab during first-line chemotherapy (yes vs no), number of standard chemotherapy courses (2-3 vs 4-6), Linear Analog Self Assessment value (≤ 7 vs > 7), and histology (predominantly squamous cell vs not predominantly squamous cell). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo observation for 6 weeks.
* Arm II: Patients undergo radiotherapy 5 days a week for 6 weeks to all sites of gross disease.

After completion of study therapy, patients are followed every 3-6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Mixed histology allowed if all components are consistent with NSCLC
  * Squamous cell histology allowed
* Stage IV disease

  * Oligometastatic disease (M1 with 1-3 metastases)

    * Patients with M1 disease that involves intrapulmonary metastases are eligible provided ≤ 40% of the total lung volume receives ≥ 20 Gy of radiotherapy
* Previously untreated disease OR achieved stable disease or partial response within 8 weeks after completion of 2-6 courses of standard platinum-based chemotherapy (administered every 3-4 weeks)
* Pleural effusion allowed provided it is minimal
* No history of or current brain metastases

  * Patients who have had up to 3 brain metastases allowed provided they have been treated with not signs of progression

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 100,00/mm^3
* Hemoglobin ≥ 9 g/dL
* WBC ≥ 2,000/mm^3
* Creatinine ≤ 2 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to undergo radiotherapy, based on radiation oncology consultation
* Willing and able to comply with study treatment
* FEV_1 ≥ 1 L
* No requirement for daily supplemental oxygen
* No second primary malignancy, except for any of the following:

  * Carcinoma in situ of the cervix
  * Nonmelanoma skin cancer
  * History of low-grade (Gleason score ≤ 6) localized prostate cancer, even if diagnosed within the past 5 years
  * Stage I breast cancer that was treated within the past 5 years
  * Other malignancy that was diagnosed and definitely treated ≥ 5 years ago with no subsequent evidence of recurrence
* No concurrent severe and/or uncontrolled medical condition, including any of the following:

  * Angina pectoris
  * Congestive heart failure within the past 3 months, unless LVEF > 40%
  * Myocardial infarction within the past 6 months
  * Cardiac arrhythmia
* No clinically significant infection
* No psychiatric illness or social situation that would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy for this cancer other than 2-6 courses of standard platinum-based chemotherapy with or without bevacizumab
* No prior radiotherapy to the treatment sites (e.g., primary lesion, clinically involved nodes, or metastatic lesions)
* No bevacizumab during and for 4 weeks after completion of radiotherapy
* No concurrent systemic chemotherapy
* No other maintenance systemic therapy during radiotherapy
* No other concurrent investigational agents for the primary neoplasm
* No concurrent intensity modulated radiotherapy
* No concurrent prophylactic nodal radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Schild, MD, Study Chair — Mayo Clinic
Locations (168):
- United States (168):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lahey Clinic Medical Center - Burlington, Burlington, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four participants were pre-registered between May 2009 and March 2010. One participant was deemed a screen failure due to eligibility reasons and 3 participants have been randomized between October 2009 and March 2010. The study was terminated prematurely on July 16, 2010 due to slow enrollment.
Pre-assignment Details: One of the randomized participants was deemed a cancel after going off study prior to receiving study treatment, thus, excluded from all analyses.
Groups:
- Arm I (No Radiation): Patients undergo observation for 6 weeks.
- Arm II (Radiation Therapy): Patients undergo radiotherapy 5 days a week for 6 weeks to all sites of gross disease.
Period: Overall Study
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who met the eligibility criteria and started the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 1 | 1
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from registration to the date of death or last follow-up
Time Frame: Time from registration to death or last follow-up (up to 5 years)
Population: Study terminated prematurely. Planned analyses was not performed. The data collected was not summarized in the data table due to the protected health information would specifically identify the study participants.
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Response Rate
Description: A confirmed tumor response was defined as a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations around 3 months apart. All participants with measurable disease (non-CR at baseline, etc.), meeting the eligibility criteria who have signed a consent form and have started the study were evaluable for response.
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the first of either death due to any cause or progression.
Time Frame: Time from registration to disease progression or death (up to 5 years)
Population: as for outcome 1
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the time from randomization to the earliest date documentation of disease progression occurs. If a patient dies without a documentation of disease progression, the patient will be considered to have had tumor progression at the time of their death unless there is sufficient documented evidence to conclude no progression occurred prior to death.
Time Frame: Time from registration to disease progression (up to 5 years)
Population: as for outcome 1
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time from the date of randomization to the date at which the patient was removed from treatment (Arm II) or no treatment (Arm I) due to progression, adverse events, or refusal.
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response
Description: Duration of response was defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status was first noted to be either a complete response (CR) or partial response (PR) to the earliest date progression was documented.
Time Frame: Up to 5 years
Population: as for outcome 1
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: All participants who met the eligibility criteria and started the study.
Arm/Group | Arm I (No Radiation) | Arm II (Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (No Radiation) (N=1) | Arm II (Radiation Therapy) (N=1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less